CLINICAL TRIAL: NCT06397131
Title: A Multicenter Study to Determine the Safety and Efficacy of NT-501 Utilizing the Medica Membrane in Macular Telangiectasia Type 2
Brief Title: A Study to Determine the Safety and Efficacy of NT-501 With MHFM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTMT-03C
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Macular Telangiectasia Type 2
Keywords: Ciliary Neurotrophic Factor; Macular Telangiectasia (MacTel) Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NT-501 CNTF Implant with Medica Hollow Fiber Membrane (MHFM) (Experimental): Participants to receive CNTF implant in one eye using MHFM.
  Interventions: Combination Product: NT-501 CNTF Implant

INTERVENTIONS:
Combination Product: NT-501 CNTF Implant — Single implantation of CNTF-secreting NT-501 hCNTF device into one eye.

SUMMARY:
This study is to determine the long-term levels of CNTF, and the clinical safety and efficacy of the NT-501 implants with the Medica Hollow Fiber Membrane (MHFM) in participants with macular telangiectasia type 2.

DETAILED DESCRIPTION:
Two parallel randomized, controlled Phase 3 clinical trials showed that placing an NT-501 in the eyes of subjects with macular telangiectasia type 2 (MacTel) provides vision benefit with an acceptable risk profile. The NT-501 device used in these Phase 3 trials has a hollow fiber membrane (HFM) which houses the CNTF producing engineered NTC-201-6A cells. The produced CNTF passes through the membrane into the vitreous cavity of the affected eye and similarly required cell nutrients pass from the vitreous cavity through the membrane to the NTC-201-6A cells. NT-501 used in the above mentioned Phase 3 studies was manufactured with the clinical HFM (referred to as CHFM) from a single sourced supplier. Another supplier of this critical HFM component of the NT-501 has been identified. This membrane will be referred to as the Medica Hollow Fiber Membrane (MHFM). Though the NT-501 product manufactured with the MHFM has the same configuration, same RPE cells, and produces CNTF levels similar to the original NT-501 product manufactured with clinical membrane (CHFM) when tested in vivo (animal model), it has not been tested in humans. The purpose of this study is to characterize the clinical safety and efficacy of NT-501 with MHFM, consistent with the clinical safety and efficacy of NT-501 with CHFM.

ELIGIBILITY:
Key Eligibility Criteria:

1. Subjects must have a positive diagnosis of MacTel with evidence of fluorescein leakage typical of MacTel and at least one of the other features that include hyperpigmentation that is outside of a 500 micron radius from the center of the fovea, retinal opacification, crystalline deposits, right-angle vessels, or inner/outer lamellar cavities seen clinically or on SD-OCT.
2. Subject must have a break in the ellipsoid zone (EZ) (area of IS/OS loss) as measured by SD-OCT between 0.16 and 2.00 millimeters squared.
3. Subject's best-corrected visual acuity (BCVA) is 54-letter score or better (20/80 or better) as measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at screening.
4. Subject must have steady fixation in the foveal or parafoveal area and sufficiently clear media for good quality retinal imaging.
5. Subject must be 21 years or older and less than 80 years of age at screening.
6. Subject or their legally authorized representative must be able to provide written informed consent to participate in the study, in accordance with the International Conference on Harmonisation Good Clinical Practices guidelines, and local regulations, before initiating any study-related procedures.

Key Exclusion Criteria:

1. Subject is medically unable to comply with study procedures or follow-up visits.
2. Subject received intravitreal steroid therapy for non-neovascular MacTel within the last 3 months.
3. Subject has ever received intravitreal anti-vascular endothelial growth factor (VEGF) therapy in the study eye OR has, within the past 3 months, received intravitreal anti-VEGF therapy in the fellow eye at randomization.
4. Subject has evidence of ocular disease other than MacTel that, in the judgment of the examining physician, may confound the diagnosis, procedures, or outcome of the study (e.g., uncontrolled glaucoma, severe non-proliferative or proliferative diabetic retinopathy, uveitis).
5. Subject has a chronic requirement (e.g., ≥ 4 weeks at a time) for ocular medications and/or has a diagnosed disease that, in the judgment of the examining physician, may be vision threatening or may affect the primary outcome. The exceptions to this exclusion criteria include artificial tears or one glaucoma medication for early or intermediate primary open-angle glaucoma.
6. Subject has evidence of intraretinal neovascularization or subretinal neovascularization (SRNV), as evidenced by hemorrhage, hard exudate, subretinal fluid or intraretinal fluid in either eye.
7. Subject has evidence of intraretinal hyperreflectivity by OCT.
8. Subject has evidence of central serous chorio-retinopathy in either eye.
9. Subject has evidence of pathologic myopia in either eye.
10. Subject has significant corneal or media opacities in either eye.
11. Subject has had a vitrectomy, penetrating keratoplasty, trabeculectomy, or trabeculoplasty.
12. Subject has any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 2, or a nuclear opacity > standard 3 as measured on the Age -Related Eye Disease Study (AREDS) clinical lens grading system.
13. Subject has undergone lens removal in the previous 3 months or YAG laser within 4 weeks.
14. Previous participation in any Neurotech MacTel clinical trial unless the participant previously consented and screened for either the NTMT-03A or NTMT-03B study and were deemed a screen failure solely due to small lesion size.
15. Subject was a participant in any other ocular related or ocular impacted clinical trial of an intervention (drug or device) within the last 6 months.
16. Subject is on chemotherapy.
17. Subject is pregnant or breastfeeding.
18. Subject has a history of malignancy that would compromise the 12-month study survival.
19. Subject with a history of ocular herpes virus in either eye.
20. Subject has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations, and outcome assessments.
21. Subject has evidence of subfoveal RPE hyperplasia.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in Ellipsoid Zone (EZ) Area Loss | Baseline through 12 months.
  Rate of change in EZ area loss as measured by en face imaging by Spectral-Domain Optical Coherence Tomography (SD-OCT) in the study eye.

SECONDARY OUTCOMES:
Safety Outcomes | Baseline to 12 months
  The number and severity of adverse events post-implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aaberg, Jr., MD, Study Chair — Neurotech Pharmaceuticals
Locations (3):
- United States (3):
  - Bay Area Retina Associates, A Medical Group, Walnut Creek, California
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Retina Consultants of Texas, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No